CLINICAL TRIAL: NCT02766998
Title: Preserved Umbilical Vein Use as Autologous Shunt Conduits in Neonatal Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Hoganson, Assistant in Cardiac Surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00021450
Record Dates: First submitted 2016-05-02; First posted 2016-05-10 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preserved umbilical vein (Experimental): Preserved umbilical vein as shunt/conduit
  Interventions: Procedure: Preserved umbilical vein as shunt/conduit

INTERVENTIONS:
Procedure: Preserved umbilical vein as shunt/conduit — All subjects will have umbilical vein harvested and stored for use in first cardiac surgery requiring shunt or conduit.

SUMMARY:
This is a prospective, single center, safety and feasibility trial to evaluate the use of autologous umbilical vein as shunts or conduits in neonatal cardiac surgery. Subjects will be identified here at the Advanced Fetal Care Center (AFCC) following diagnosis of congenital heart disease (CHD) with single ventricle physiology of the fetus via fetal echocardiogram. At time of cesarean section or vaginal delivery, umbilical cord will be harvested in a sterile fashion and the umbilical vein will be dissected free and preserved until first clinically indicated Stage I palliative procedure between day 3 and 7 of life. Subjects will be followed until their Stage II palliative procedure.

ELIGIBILITY:
Inclusion Criteria:

* All fetal diagnoses of complex congenital heart disease diagnosed by fetal echocardiogram requiring cardiac repair with Blalock-Taussig Shunt or Right Ventricle to Pulmonary Artery conduit will be eligible.
* This includes all pre-natal diagnoses of any single ventricle circulation physiology (SVP).
* Subjects being delivered via cesarean section or vaginally at Brigham and Women's Hospital will be considered.

Exclusion Criteria:

* meconium at delivery
* symptomatic Group B Streptococcus (GBS) positive mothers
* mothers with chorioamnionitis
* Hepatitis B or C positive mothers
* HIV positive mothers.
* If unable to collect viable cord on the day of delivery of already enrolled subjects, the subject will be removed from the study on day of birth.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Absense of primary serious adverse events | from time of insertion to time of Stage II procedure, approximately 6 months
  Primary SAEs are defined as:
  * Bleeding from shunt/conduit requiring intervention (either medical or surgical)
  * Shunt/conduit thrombosis
  * Shunt/conduit infection with positive culture of preservative solution or positive clinical culture following implantation of umbilical vein
  * Aneurysm of shunt/conduit

CONTACTS AND LOCATIONS:
Overall Officials: Sitaram Emani, MD, Principal Investigator — Cardiovascular Surgeon
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States